CLINICAL TRIAL: NCT03660696
Title: Qatar Cardiovascular Biorepository-AF (QCBio-AF) Study
Brief Title: Qatar Cardiovascular Biorepository of AF Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-17-001
Record Dates: First submitted 2018-07-24; First posted 2018-09-06 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: None Retained — patients and family members with AF to enable subsequent clinical, molecular, and genetic studies. We outline here the rationale for studies that will utilize this resource, as well as specific hypotheses that will be evaluated and approaches that will be undertaken
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Qatar Cardiovascular Biorepsoitory-AF (QCBio-AF) of plasma and DNA of Qatari patients with atrial fibrillation (AF) is to establish. AF cases will include patients with acute and chronic AF identified in the Heart Hospital (HH) arrhythmia clinics and Emergency Room (ER). Controls will include blood donors who have no history of AF. Such a resource will enable validation of biomarkers to assess AF risk, response to therapy, and prognosis. QCBio-AF will also allow genomic, marker and proteomic studies of AF and response to drug therapy (pharmacogenetics and pharmacoproteomics). This study will accomplish the following specific aims: Aim 1: Establish a DNA and plasma biorepository (QCBio-AF) of 300 Qatari AF cases and Family members to enable investigation of genomic and proteomic biomarkers for early detection and prognostication and to identify new targets for drug development. Aim 2: Annotate the biorepository of with 1) demographic, laboratory, and clinical variables derived from the EMR using electronic phenotyping algorithms, and 2) detailed information regarding history of cardiovascular diseases and risk factors derived from patient surveys. Aim 3: Develop processes to promote use of the biorepository by Qatari investigators by facilitating access to the biorepository for biomarker research, while maintaining the highest ethical standards with emphasis on patient confidentiality and stewardship of the biospecimens. Timeline. Following IRB approval, the intended collection period will be over 12 months where 300 Qatari patients with AF and their immediate families will be recruited. Significance: Although atrial fibrillation (AF) is reaching epidemic proportions in the aging U.S. and European populations, the worldwide burden of AF in non-white populations is unknown. Furthermore, a substantial proportion of AF in the population is not explained by traditional risk factors. There is increasing evidence that susceptibility to AF is not only determined by underlying etiologic risk factors but also ethnicity with AF occurring more frequently in white than in non-white populations. While reasons for this ethnic variability are unknown, studies have shown that both common and rare genetic variants increase susceptibility to AF in an individual in the presence of ethnic-specific risk factors.

DETAILED DESCRIPTION:
Atrial Fibrillation Epidemic and the Need for Improved Therapies: Atrial fibrillation (AF) has become a disease of global epidemic proportions due to the burgeoning population of elderly individuals. The global burden of AF was recently estimated at 33.5 million with progressive increases in incidence, prevalence and AF-related mortality having major implications for healthcare costs and public health policy. This study also highlighted regional variation in AF burden between developed versus developing countries. The number of persons in the U.S. with AF by the year 2050 is projected to exceed 16 million. The socioeconomic impacts of AF are substantial, as are the consequences of frequent visits to the emergency room (ER) and hospitalizations, chronic disease management and loss of productivity. Moreover, managing patients with AF remains challenging. Despite recent advances in catheter-based and surgical treatments, antiarrhythmic drugs (AADs) remain the mainstay of treatment for patients with symptomatic AF. However, membrane active drugs are incompletely and unpredictably effective and can be proarrhythmic. Furthermore, the selection of an AAD for an individual patient is based not only on efficacy as on minimizing the risk of adverse effects. The limited success of AADs in maintaining sinus rhythm is related in part to the heterogeneity of the underlying substrate, poor understanding of the pathophysiology of AF and our failure to target therapy to underlying mechanisms. Thus, an overarching goal of this proposal is to create and utilize a clinical and genetic database for AF to examine the role of novel and established risk factors for AF in diverse ethnic populations and determine the role of common AF susceptibility loci in two ethnic groups and examine gene-environment interactions between ethnic specific risk factors and AF.

Genetic Epidemiology of AF, in 1943, first report of familial AF in three brothers with early onset AF published. Since then many epidemiologic studies have shown that AF is heritable especially the form of AF that occurs without underlying cardiac or systemic disease - previously termed lone but is now designated as early onset AF. As the heritability of AF has been estimated to be 62%, there is a substantial genetic component to the arrhythmia. While some of loci influencing this estimate may be pleiotropic and related to other risk factors such as hypertension and diabetes that are also highly heritable, there are also several discovered and likely many undiscovered genetic risk factors that are primary determinants of early onset AF. Many genes and several AF loci have now been identified for Mendelian forms of early onset AF. In 1997, Brugada and colleagues identified the first AF locus on chr10q22; since then four other loci have been identified, including a new locus on chr5p15 identified by us that was associated with a prolonged P-wave duration. In addition, linkage analyses have identified individual mutations in several familial AF kindreds. The first AF gene (KCNQ1), identified in 2003, encodes a cardiac potassium channel current (IKs). This discovery was followed by the identification of other potassium and cardiac ion channels important in the pathophysiology of AF. The first non-ion channel AF gene (natriuretic peptide precursor A [NPPA]), was identified by linkage analysis and a positional cloning approach and encodes for atrial natriuretic peptide (ANP).

With the discovery of KCNQ1 as an AF gene, investigators then applied a candidate gene approach and identified many more rare 'private' genetic variants in other cardiac ion channel genes in familial AF kindreds. In 2007, Otway and colleagues identified a KCNQ1 mutation (R14C) in one family with familial AF. When the mutation was expressed in a heterologous expression system, the IKs current amplitude at baseline was unchanged but demonstrated marked increase compared to wild-type (WT) channels when exposed to hypotonic solution. Importantly, only those subjects with left atrial (LA) dilatation developed AF. These findings and Vanderbilt data showing that penetrance of rare AF-associated variants is modulated by common AF risk alleles at the chr4q25 locus support the concept of a two-hit genetic model for the development of AF. Mutations in genes encoding connexins, proteins important in transmitting electrical activity between cardiac myocytes, have also been identified stemming from early work in mice with null alleles for GJA5, encoding mutations in several familial AF kindreds. The first AF gene (KCNQ1), identified in 2003, encodes a cardiac potassium channel current (IKs). This discovery was followed by the identification of other potassium and cardiac ion channels important in the pathophysiology of AF. The first non-ion channel AF gene (natriuretic peptide precursor A [NPPA]), was identified by linkage analysis and a positional cloning approach and encodes for atrial natriuretic peptide (ANP).

Epidemiology of AF in Qatar: The burden of AF in populations of Middle Eastern Arabs remains unknown. Researchers explored the etiology and pattern of AF in Middle Eastern Arabs and South Asians living in Qatar using the CCS Registry at HMC26 and showed that, in this population, AF is more common in those that are older, have a history of HTN, CHF, DM and valvular heart disease. Furthermore, they showed that the incidence of AF in Middle Eastern Arab patients was significantly higher than in South Asians (12% vs. 8%) and this was mostly due to older age, a greater prevalence of HTN, and DM in the Arabs. The Registry was also used to compare the clinical demographics, and management of AF in Middle Eastern Arab in Qatar. Over 2800 Arabs and 500 South Asians were admitted for evaluation and management of AF over the 20-year period. Middle Eastern Arabs with AF were older, and had a greater prevalence of HTN, DM, chronic renal insufficient and hyperlipidemia. In contrast, South Asians were more likely to have acute coronary syndromes and a history of valvular heart disease. Importantly the in-hospital mortality rate was higher in Arabs than South Asians but the stroke rates were comparable. These studies highlight the differential impact of traditional risk factors on the development of AF in Middle eastern Arabs.

Identification of probands and families with early-onset AF in Qatar: Two Middle Eastern Arab families have been identified with early-onset AF. In one family, three family members besides the proband presented with highly symptomatic AF at age <40 years. In the second family, six family members have presented with early-onset AF. These findings are very preliminary evaluations and upon approval of the submitted protocol by the IRB Ethics Committee, further evaluations of these two families will take place.

Participant recruitment and enrollment: Patients who are over the age of 18 years presenting with early-onset AF from cardiology clinics, the ER and in-patient services from the HMC network of hospitals (Hamad General Hospital, Hamad Heart Hospital, Al-Khor Hospital, Cuban Hospital, and Al-Wakra Hospital). The HMC hospital network provides both outpatient and in-patient cardiology services for all Qatar residents, and >95% of all cardiac patients in the country are treated at these hospitals, including patients with acute cardiac conditions, representing essentially a population-based cohort for identification and selection of AF patients and a control cohort of non-AF cardiology patients for the genetic studies. These participants will comprise two broad ethnic groups that have not been adequately studied previously, defined as: Qatari and other Middle Eastern Arabs. A diagnosis of AF will be confirmed when an ECG shows AF during the index hospitalization/ER visit showing AF. Patients with a history of AF only in the setting of cardiac surgery will be excluded from this study.

For this proposal, only family members of Qatari Middle Eastern Arab patient with early onset (≤60 years of age) AF will be targeted for recruitment. In 2016, over 600 patients with AF were seen in the Hamad General Hospital ER and over 400 patients were seen by Dr. Nidal Assad (LPI) in the Arrhythmia Clinic at the Hamad Heart Hospital. Approximately 30% of these patients presented with early-onset AF. A projected annual growth of over 20% in new patients with AF will not only increase the likelihood of meeting our target recruitment but will also significantly improve our chances of identifying large kindreds with familial AF. At the same network of hospitals during the same time period, It will identify a cohort of cardiology patients without AF to be followed prospectively and to serve as a comparison group for genetic analyses. This control cohort will be a representative sample of the population of cardiology patients who do not have AF, which is already available from another completed cardiology biorepository. Patients will not be enrolled if major difficulties with follow-up are anticipated, for example, patients with no valid residency permit or those planning to leave the country before the next planned follow-up visit.

Subject Population(s) Total number of QCBio-AF participants: 300 Age range of participants: 18 yrs and above Targeted number of males: 150 Targeted number of females: 150 A informed consent will be indicated to recruit patients who may be eligible for the study.

Participant Identification, Inclusion/Exclusion Criteria, and Recruitment Patients will be identified through Hamad Medical Corporation (HMC) Heart Hospital (HH) Arrhythmia and General Cardiology Clinics and the Emergency Department will be approached for inclusion in the study. A detailed family history and a DNA sample will then be obtained by the principal investigator or a research coordinator, following written informed consent under a protocol approved by the Institutional Review Board of HMC. Upon identification of a patient with a family history of AF, relatives will be contacted by the by the principal investigator or a research coordinator. Once this is obtained, outside medical records will be requested.

Identify the criteria for inclusion and exclusion and explain the procedures that will be used to determine eligibility:

Specimen Collection for the main study:

Blood drawing (indicate total amount drawn for research purposes): 25 cc x 1 (one-time only).

Other specimens (describe the type of specimen and frequency of collection): None Study-specific questionnaires will be conducted at enrollment, and when appropriate and available, collected at the subjects' six-month and 12-month scheduled clinic visits. The questionnaires will take approximately take 10 minutes to complete. These are only applicable to adult patients.

The baseline, 6-month, and 12-month questionnaires and other information from the medical record will be collected at regularly scheduled clinic visits on study-specific source documentation to later be transcribed onto SPSS with only the subject's study-specific code ID/number assigned to the data.

The ECG, ECHO, and Holter monitoring will be performed (or will have already been performed) as part of the subjects' clinically indicated treatment/management for their AF. Family members asked to participate in the study who do not have a documented history of AF will not have the ECG, ECHO, and Holter monitoring performed because it is not clinically indicated. Family members who are not part of the UIC medical system and have had an ECG, ECHO, and/or Holter monitoring performed at outside facilities will be asked to provide this information for research purposes only.

The creation of a Qatar Cardiovascular Biorepsoitory-AF (QCBio-AF): a resource that will collect and store clinical, demographic, blood and DNA samples from patients and family members with AF to enable subsequent clinical, molecular, and genetic studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years
2. History of AF and without
3. Atrial flutter by ECG, ECHO or Holter monitor event recorder
4. Willing to give written informed consent.

Exclusion Criteria:

1. AF or atrial flutter associated with cardiac surgery
2. Pregnant females (at the baseline visit) and prisoners.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Qatari subjects must have a documented history of AF or atrial flutter by ECG, ECHO, and or Holter monitor event recorder. Subjects' family members approached for the study may or may not have a documented history AF.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of KCNQ1 Gene expression in AF | One year
  Establish a DNA and plasma biorepository (QCBio-AF) of 300 Qatari AF cases and Family members to enable investigation of genomic and proteomic biomarkers for early detection and prognostication and to identify new targets for drug development
Incidence of AF in diverse ethnic population | One year
  Risk factors for AF in diverse ethnic population

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Hospital, Hamad Medical Coorporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chugh SS, Havmoeller R, Narayanan K, Singh D, Rienstra M, Benjamin EJ, Gillum RF, Kim YH, McAnulty JH Jr, Zheng ZJ, Forouzanfar MH, Naghavi M, Mensah GA, Ezzati M, Murray CJ. Worldwide epidemiology of atrial fibrillation: a Global Burden of Disease 2010 Study. Circulation. 2014 Feb 25;129(8):837-47. doi: 10.1161/CIRCULATIONAHA.113.005119. Epub 2013 Dec 17. PMID 24345399
- [Result] Stewart S, Murphy NF, Walker A, McGuire A, McMurray JJ. Cost of an emerging epidemic: an economic analysis of atrial fibrillation in the UK. Heart. 2004 Mar;90(3):286-92. doi: 10.1136/hrt.2002.008748. PMID 14966048
- [Result] Bruggenjurgen B, Rossnagel K, Roll S, Andersson FL, Selim D, Muller-Nordhorn J, Nolte CH, Jungehulsing GJ, Villringer A, Willich SN. The impact of atrial fibrillation on the cost of stroke: the berlin acute stroke study. Value Health. 2007 Mar-Apr;10(2):137-43. doi: 10.1111/j.1524-4733.2006.00160.x. PMID 17391422
- [Result] Fox CS, Parise H, D'Agostino RB Sr, Lloyd-Jones DM, Vasan RS, Wang TJ, Levy D, Wolf PA, Benjamin EJ. Parental atrial fibrillation as a risk factor for atrial fibrillation in offspring. JAMA. 2004 Jun 16;291(23):2851-5. doi: 10.1001/jama.291.23.2851. PMID 15199036
- [Result] Arnar DO, Thorvaldsson S, Manolio TA, Thorgeirsson G, Kristjansson K, Hakonarson H, Stefansson K. Familial aggregation of atrial fibrillation in Iceland. Eur Heart J. 2006 Mar;27(6):708-12. doi: 10.1093/eurheartj/ehi727. Epub 2006 Jan 20. PMID 16428254
- [Result] Christophersen IE, Ravn LS, Budtz-Joergensen E, Skytthe A, Haunsoe S, Svendsen JH, Christensen K. Familial aggregation of atrial fibrillation: a study in Danish twins. Circ Arrhythm Electrophysiol. 2009 Aug;2(4):378-83. doi: 10.1161/CIRCEP.108.786665. Epub 2009 Apr 23. PMID 19808493
- [Result] Salam AM, AlBinali HA, Al-Mulla AW, Singh R, Al Suwaidi J. Secular trends, treatments, and outcomes of Middle Eastern Arab and South Asian patients hospitalized with atrial fibrillation: insights from a 20-year registry in Qatar (1991-2010). Angiology. 2013 Oct;64(7):498-504. doi: 10.1177/0003319712460332. Epub 2012 Oct 1. PMID 23028177
- [Result] Salam AM, AlBinali HA, Al-Mulla AW, Asaad N, Singh R, Al-Qahtani A, Al Suwaidi J. Women hospitalized with atrial fibrillation: gender differences, trends and outcome from a 20-year registry in a Middle Eastern country (1991-2010). Int J Cardiol. 2013 Sep 30;168(2):975-80. doi: 10.1016/j.ijcard.2012.10.041. Epub 2012 Nov 15. PMID 23159409
- [Result] Salam AM, AlBinali HA, Al-Sulaiti EM, Al-Mulla AW, Singh R, Al Suwaidi J. Effect of age on treatment, trends and outcome of patients hospitalized with atrial fibrillation: insights from a 20-years registry in a Middle-Eastern country (1991-2010). Aging Clin Exp Res. 2012 Dec;24(6):682-90. doi: 10.3275/8757. Epub 2012 Nov 26. PMID 23211770